CLINICAL TRIAL: NCT02570074
Title: Phase I Study to Evaluate Pharmacokinetics, Pharmacodynamics and Safety/Tolerability of Two Dosing Regimens of Oral Fosfomycin Tromethamine in Healthy Adult Participants
Brief Title: PK/PD and Safety/Tolerability of Two Dosing Regimens of Oral Fosfomycin Tromethamine in Healthy Adults
Acronym: PROOF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vance Fowler, M.D. (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Vance Fowler, M.D., Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00066102; 1UM1AI104681-01 (NIH)
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Fosfomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fosfomycin - 3 doses QoD/7 doses QD (Experimental): Fosfomycin given as a 3 gm dose, every other day for 3 doses, followed by 3 gm dose, once a day for 7 doses.
  Interventions: Drug: Fosfomycin
- Fosfomycin - 7 doses QD/3 doses QoD (Experimental): Fosfomycin given as a 3 gm dose, once a day for 7 doses, followed by 3 gm dose, every other day for 3 doses.
  Interventions: Drug: Fosfomycin

INTERVENTIONS:
Drug: Fosfomycin — Broad spectrum antibiotic

SUMMARY:
Oral dosage regimens for fosfomycin tromethamine (Monurol™) are not established for the treatment of cUTI. The most common and recommended adult dosage regimen in the literature is a single-dose sachet containing the equivalent of 3 grams of fosfomycin administered every other day (QOD) for a total of three doses.

There are a myriad of different oral fosfomycin dosing regimens currently being used in clinical practice, including up to 3 grams orally twice daily for 7-21 days, but these regimens are not based on solid pharmacokinetic, pharmacodynamic or safety rationale. Initial pharmacokinetic studies performed with oral fosfomycin tromethamine primarily examined single dose regimens and did not use modern day bioanalytical or pharmacokinetic techniques. As the use of fosfomycin becomes more pervasive in concordance with the increase in multidrug resistant pathogens, further pharmacokinetic and safety data are needed for more intensive dosing regimens to support its continued use.

The rationale of this study is that oral fosfomycin tromethamine requires a modern pharmacokinetic-pharmacodynamic study to identify alternative oral dosage regimens that are appropriate and safe. This study provided safety/tolerability and clinical pharmacology information regarding two oral dosing regimens that may have application to treat various types of infections involving resistant pathogens or when other oral antibacterial options are not available.

DETAILED DESCRIPTION:
The study was designed as a randomized, two-way crossover trial involving up to 24 randomized participants with an anticipated drop-out rate no higher than 25% to give a total of 18 evaluable healthy adult participants. The study was fully explained to each participant, informed consent was obtained, and an IRB-approved informed consent form was signed before any study procedures were initiated. All participants underwent screening assessments within 30 days prior to the initial dosing to determine their eligibility for enrollment into the study. All participants met the inclusion and exclusion criteria and underwent screening procedures that included a complete medical history, physical examination, assessment of clinical laboratory parameters (chemistry and hematology), ECG, and pregnancy test (females of child bearing potential only).

Randomization was stratified by gender, using permuted blocks. Within each gender, eligible participants were randomized with equal probability to one of the 2 treatment sequences shown in Table 3. According to the sequence to which the participant was randomized, the participant initially received one of two oral dosage regimens of fosfomycin: 3 g every other day x 3 doses or 3 g once-daily x 7 doses. After completion of the initial dosing regimen each participant was crossed over to receive the other dosing regimen. There was a minimum 5-day, and a recommended maximum 14-day, washout period prior to starting the next dosing regimen. Blood and urine samples were collected throughout the study as well as detailed drug administration and adverse event data for each participant.

Fosfomycin tromethamine sachet (Monurol™) was used in this study. Each participant was instructed how to stir and dissolve the single-dose sachet into 3 to 4 ounces of water, and take each dose immediately after dissolving in water. Compliance was assessed by participant interviews (every 2 days) and counting of empty of sachets.

Participants reported to the outpatient study center on Day -30 to -1 for study criteria review, clinical assessment, and blood collection for screening laboratory tests prior to fosfomycin administration. Each participant participated in the study up to 120 days (i.e., screening visit; day -1 for clinical assessment and blood collection; days 1-7 for fosfomycin administration and sample collection period; and day 8-10 for follow-up assessment; crossed over to receive the other dosing regimen and schedule of events.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is healthy as judged by the site investigator with no clinically significant abnormality identified on a medical evaluation including history, physical examination, laboratory tests, blood pressure, and heart rate.
2. Male and female participants between 18 to 55 years old.
3. Female participants of childbearing potential (not surgically sterilized and between menarche and one-year post-menopause) must have a negative pregnancy test at the time of enrollment and must agree to use appropriate contraception for as long as they are taking the study drug and for 1 month afterwards. During the screening visit, participants will be instructed to use a second reliable method of birth control in accordance with the protocol during the study and for one month following. Medically acceptable contraceptives include:

   * Surgical sterilization (such as a tubal ligation or hysterectomy)
   * Approved hormonal contraceptives (such as birth control pills, patches, implants or injections)
   * Barrier methods (such as a condom or diaphragm) used with a spermicide, or
   * An intrauterine device (IUD). i. NOTE: Contraceptive measures such as Plan B™, sold for emergency use after unprotected sex, are not acceptable methods for routine use.
4. Nonsmokers defined as abstinence from cigarette smoking for the previous 6 months before enrollment into the study.
5. Provide a signed and dated written informed consent prior to any study-specific procedures (including screening procedures).
6. Body weight ≥50 kg
7. Body mass index (BMI) 18.5-29.9 kg/m2

Exclusion Criteria:

1. History of significant hypersensitivity reaction or intolerance to fosfomycin tromethamine that in the opinion of the site investigator, contraindicates participation in the study. In addition, if heparin is used during pharmacokinetic sampling, participants with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
2. History of significant cardiac, neurological, thyroid, muscular, or immune disorder.
3. Any laboratory abnormality grade 2 or higher as defined according to the U.S. Department of Health and Human Services common terminology criteria for AEs (CTCAE).26
4. Estimated creatinine clearance (CLCR) <60 ml/minute as determined by Cockcroft-Gault equation
5. Positive serum pregnancy test.
6. Currently breast feeding.
7. History of alcohol or substance abuse or dependence within 6 months of the screening: History of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men. 1 drink is equivalent to 12g alcohol = 5 oz (150 mL) of wine or 12 oz (360 mL) of beer or 1.5 oz (45 mL) of 80 proof distilled spirits.
8. The use of prescription (except birth control pills or hormone replacement in females) or non-prescription drugs, including herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of site investigator the medication will not interfere with the study procedures or compromise participant safety.
9. The participant has participated in a clinical trial and has received a drug or a new chemical entity within 30 days prior to the first dose of study medication.
10. Participants who have donated blood to the extent where participation in the study would result in excess of 500 mL blood donated within a 56 day period.
11. Those who, in the opinion of the site investigator, have a risk of non-compliance with study procedures.
12. QTc interval with Fredericia correction >450ms or any other clinically relevant ECG abnormalities

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vance Fowler, MD, Principal Investigator — Duke University
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wenzler E, Meyer KM, Bleasdale SC, Sikka M, Mendes RE, Bunnell KL, Finnemeyer M, Rosenkranz SL, Danziger LH, Rodvold KA. Ex Vivo Urinary Bactericidal Activity and Urinary Pharmacodynamics of Fosfomycin after Two Repeated Dosing Regimens of Oral Fosfomycin Tromethamine in Healthy Adult Subjects. Antimicrob Agents Chemother. 2020 Jan 27;64(2):e02102-19. doi: 10.1128/AAC.02102-19. Print 2020 Jan 27. PMID 31767717
- [Derived] Wenzler E, Bleasdale SC, Sikka M, Bunnell KL, Finnemeyer M, Rosenkranz SL, Danziger LH, Rodvold KA; Antibacterial Resistance Leadership Group. Phase I Study To Evaluate the Pharmacokinetics, Safety, and Tolerability of Two Dosing Regimens of Oral Fosfomycin Tromethamine in Healthy Adult Participants. Antimicrob Agents Chemother. 2018 Jul 27;62(8):e00464-18. doi: 10.1128/AAC.00464-18. Print 2018 Aug. PMID 29891606

RESULTS

PARTICIPANT FLOW:
Period: Period 1 (First Dosing Regimen)
Arm/Group | Fosfomycin - 3 Doses QoD/7 Doses QD | Fosfomycin - 7 Doses QD/3 Doses QoD
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0
Period: Period 2 (Second Dosing Regimen)
Arm/Group | Fosfomycin - 3 Doses QoD/7 Doses QD | Fosfomycin - 7 Doses QD/3 Doses QoD
Started | 9 | 10
Completed | 8 | 10
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fosfomycin - 3 Doses QoD/7 Doses QD | Fosfomycin - 7 Doses QD/3 Doses QoD | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [25 to 29] | 27 [25 to 28] | 27 [25 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 7 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
Weight [Mean (Standard Deviation); unit: kilogram] | 75.3 (12.3) | 76.0 (10.9) | 75.7 (11.3)
Entry site - University of Illinois Chicago [Number; unit: participants] | 9 | 10 | 19
Height [Mean (Standard Deviation); unit: centimeter] | 173.2 (12.0) | 173.8 (7.9) | 173.6 (9.7)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.0 (2.5) | 24.9 (2.4) | 24.9 (2.4)
Estimated creatinine clearance [Mean (Standard Deviation); unit: mL/min] | 105.0 (14.6) | 113.7 (23.0) | 109.6 (19.4)
QTC Interval [Mean (Standard Deviation); unit: milliseconds] — Average of 3 measures
  milliseconds | 402.8 (19.7) | 405.2 (17.2) | 404.1 (17.9)

OUTCOME MEASURES:

1. Primary Outcome: Number (%) of Grade 2 or Higher AEs Regardless of Relationship to Study Drug
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Fosfomycin - 3 Doses QoD Regimen; Fosfomycin - 7 Doses QD Regimen: The number of all AE is summarized by treatment but not sequence. The total number of subjects analyzed is 19.
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Participants | 1 | 3

2. Primary Outcome: Day 1: Plasma PK Concentrations [mg/L]
Description: Day 1 mean and standard deviation plasma concentrations [mg/L] at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours from dose
Time Frame: Day 1: 0, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours from dose
Population: Please note that one person did not complete the Fosfomycin 3 doses QoD regimen.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Fosfomycin - 3 Doses QoD: The analysis is by Dosing Regimen
- Fosfomycin - 7 Doses QD: The analysis is by by dosing regimen
Arm/Group | Fosfomycin - 3 Doses QoD | Fosfomycin - 7 Doses QD
Number analyzed (Participants) | 18 | 18
mg/L
  0 hours | 0.08 (0.36) | 0 (0)
  1 hour | 16.61 (5.44) | 15.90 (6.70)
  1.5 hours | 22.20 (7.98) | 21.35 (7.17)
  2 hours | 23.36 (7.04) | 22.12 (6.34)
  3 hours | 18.72 (5.13) | 17.86 (4.67)
  4 hours | 14.08 (4.00) | 13.53 (3.87)
  6 hours | 9.11 (2.38) | 8.43 (2.38)
  8 hours | 6.08 (1.48) | 5.69 (1.57)
  12 hours | 3.43 (1.01) | 3.19 (1.28)
  24 hours | 0.88 (0.59) | 1.33 (2.70)

3. Primary Outcome: Day 5: Plasma PK Concentrations [mg/L]
Description: Day 5 mean and standard deviation plasma concentrations [mg/L] at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours from dose
Time Frame: Day 5: 0, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours from dose
Population: Please note that one person did not complete the Fosfomycin 3 doses QoD regimen.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Fosfomycin - 3 Doses QoD | Fosfomycin - 7 Doses QD
Number analyzed (Participants) | 18 | 18
mg/L
  0 hours | 0.23 (0.37) | 1.33 (1.12)
  1 hour | 16.29 (6.23) | 16.81 (4.27)
  1.5 hours | 21.21 (6.91) | 22.07 (5.02)
  2 hours | 22.48 (6.44) | 23.37 (5.71)
  3 hours | 19.38 (5.34) | 19.45 (5.10)
  4 hours | 14.98 (4.82) | 15.12 (4.27)
  6 hours | 9.78 (3.08) | 9.91 (2.74)
  8 hours | 6.47 (1.95) | 6.93 (1.96)
  12 hours | 3.71 (1.31) | 4.02 (1.61)
  24 hours | 0.82 (0.40) | 1.12 (1.07)

4. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: To estimate the fosfomycin pharmacokinetic parameter maximum plasma concentration (Cmax) at steady-state for orally-dosed fosfomycin tromethamine in healthy adult participants
Time Frame: 24 hours
Population: Please note that one person did not complete the Fosfomycin 3 doses QoD regimen.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Fosfomycin - 3 Doses QoD Regimen; Fosfomycin - 7 Doses QD Regimen: The analysis is by dosing regimen.
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 18 | 18
mg/L
  Day 1 | 23.79 (7.48) | 23.47 (6.62)
  Day 5 | 24.41 (6.23) | 23.75 (5.61)

5. Primary Outcome: Day 1: Area Under the Concentration Time Curve (AUC 0-infinity)
Description: To estimate the fosfomycin pharmacokinetic parameter area-under-the-plasma concentration-time curve (AUC 0-infinity) at steady-state for orally-dosed fosfomycin tromethamine in healthy adult participants
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg*hour/L
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 18 | 18
mg*hour/L | 148.57 (35.57) | 176.44 (176.96)

6. Primary Outcome: Day 5: Area Under the Concentration Time Curve (AUC Tau-infinity)
Description: To estimate the fosfomycin pharmacokinetic parameter area-under-the-plasma concentration-time curve (AUC 0-tau) at steady-state for orally-dosed fosfomycin tromethamine in healthy adult participants
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg*hours/L
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 18 | 18
mg*hours/L | 151.60 (35.61) | 156.62 (42.52)

7. Primary Outcome: Number of Subjects Who Prematurely Discontinue Study Drug
Time Frame: Dosing period: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Fosfomycin - 3 Doses QoD: Fosfomycin given as a 3 gm dose, every other day for 3 doses.
  Fosfomycin: Broad spectrum antibiotic
- Fosfomycin - 7 Doses QD: Fosfomycin given as a 3 gm dose, once a day for 7 doses
  Fosfomycin: Broad spectrum antibiotic
Arm/Group | Fosfomycin - 3 Doses QoD | Fosfomycin - 7 Doses QD
Number analyzed (Participants) | 19 | 18
Participants | 1 | 0

8. Secondary Outcome: Total Body Clearance (CL)
Time Frame: Pooled over 24 hours: Day 1
Measure: Mean (Standard Deviation); unit: L/h
Groups:
- Fosfomycin - 3 Doses QoD Regimen; Fosfomycin - 7 Doses QD Regimen: The number of all AE is summarized by regimen but not sequence. The total number of subjects analyzed is 18.
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 18 | 18
L/h | 21.62 (6.79) | 21.96 (6.51)

9. Secondary Outcome: Apparent Volume of Distribution (Vss)
Time Frame: Pooled over 24 hours at Day 1 and Day 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Fosfomycin - 3 Doses QoD | Fosfomycin - 7 Doses QD
Number analyzed (Participants) | 18 | 18
L
  Day 1 | 172.25 (70.41) | 143.97 (55.31)
  Day 5 | 140.57 (67.94) | 146.68 (67.64)

10. Secondary Outcome: Elimination Rate Constant (z)
Time Frame: Pooled over 24 hours at Day 1 and Day 5
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Fosfomycin - 3 Doses QoD | Fosfomycin - 7 Doses QD
Number analyzed (Participants) | 18 | 18
1/h
  Day 1 | 0.13 (0.04) | 0.17 (0.06)
  Day 5 | 0.16 (0.04) | 0.16 (0.05)

11. Secondary Outcome: Elimination Half-life (t½)
Time Frame: Pooled over 24 hours at Day 1 and Day 5
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Fosfomycin - 3 Doses QoD | Fosfomycin - 7 Doses QD
Number analyzed (Participants) | 18 | 18
h
  Day 1 | 5.56 (1.54) | 5.90 (7.16)
  Day 5 | 7.53 (4.09) | 7.31 (3.46)

12. Secondary Outcome: Renal Clearance (CLR)
Time Frame: Pooled over 24 hours at Day 1 and Day 5
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Fosfomycin - 3 Doses QoD | Fosfomycin - 7 Doses QD
Number analyzed (Participants) | 18 | 18
L/h
  Day 1 | 7.10 (3.64) | 8.09 (5.60)
  Day 5 | 7.53 (4.09) | 7.31 (3.46)

13. Secondary Outcome: Amount Excreted in the Urine (Ae)
Time Frame: Pooled over 24 hours at Day 1 and Day 5
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 18 | 18
mg
  Day 1 | 1047.05 (710.53) | 1102.34 (772.67)
  Day 5 | 1177.24 (790.76) | 1161.57 (718.09)

14. Secondary Outcome: Urinary Bactericidal (UBT) Titers for E. Coli ATCC 25922
Description: UBT for E.coli ATCC 25922
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: Reciprocal Titers
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Reciprocal Titers
  Day 1, >0 to 4 hr | 4 [1 to 16] | 8 [0 to 16]
  Day 1, 4 to 8 hr | 8 [2 to 32] | 4.5 [0 to 16]
  Day 1, 8 to 12 hr | 4 [0 to 8] | 3 [1 to 8]
  Day 1, 12 to 24 hr | 4 [1 to 8] | 6 [2 to 8]
  Day 5, >0 to 4 hr | 4 [1 to 16] | 4 [1 to 16]
  Day 5, 4 to 8 hr | 12 [1 to 32] | 12 [1 to 32]
  Day 5, 8 to 12 hr | 6 [1 to 16] | 6 [1 to 16]
  Day 5, 12 to 24 hr | 4 [1 to 8] | 4 [1 to 8]

15. Secondary Outcome: Urinary Bactericidal Kinetics (UBK)
Time Frame: 3 months
Population: Data not collected.
Arm/Group | Fosfomycin - 3 Doses QoD/7 Doses QD | Fosfomycin - 7 Doses QD/3 Doses QoD
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Urine Fosfomycin Concentrations [mg/L]
Description: Urine Fosfomycin concentrations [mg/L]
Time Frame: Day 1: 24 hours
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Fosfomycin - 3 Doses QoD | Fosfomycin - 7 Doses QD
Number analyzed (Participants) | 18 | 18
mg/L
  Pre-dose | 0 (0) | 0 (0)
  0-4 hours post-Dose | 471.71 (423.10) | 563.55 (665.94)
  4-8 hours post-dose | 584.23 (348.46) | 402.90 (367.31)
  8-12 hours post dose | 201.99 (119.22) | 228.13 (163.30)
  12-24 hours post dose | 202.73 (149.08) | 175.13 (102.21)

17. Secondary Outcome: UBT-time Curve (AUBT24)
Description: For pathogens E. coli ATCC 25922, E. coli ATCC BAA-2323, K. pneumoniae ATCC 33495, K. pneumoniae ATCC 700603 and P. mirabilis ATCC 35659
Time Frame: 24 hours at Day 1 and Day 5
Measure: Mean (Standard Deviation); unit: titers * hours
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
titers * hours
  E. coli ATCC 25922, Day 1 | 175.37 (174.30) | 158.67 (199.12)
  E. coli ATCC 25922, Day 5 | 202.53 (218.71) | 196.67 (214.84)
  E. coli ATCC BAA-2323, Day 1 | 139.47 (140.45) | 121.56 (145.88)
  E. coli ATCC BAA-2323, Day 5 | 198.84 (219.90) | 156.33 (172.96)
  K. pneumoniae ATCC 33495, Day 1 | 15.68 (17.75) | 11.67 (11.95)
  K. pneumoniae ATCC 33495, Day 5 | 20.63 (19.11) | 17.44 (16.13)
  K. pneumoniae ATCC 700603, Day 1 | 10.32 (8.23) | 4.56 (7.02)
  K. pneumoniae ATCC 700603, Day 5 | 12.42 (8.83) | 9.89 (6.74)
  P. Mirabilis ATCC 35659, Day 1 | 96.53 (135.80) | 53.78 (70.75)
  P. Mirabilis ATCC 35659, Day 5 | 96.95 (148.42) | 90.33 (146.85)

18. Secondary Outcome: Urine Fosfomycin Concentrations [mg/L]
Description: Urine Fosfomycin concentrations [mg/L]
Time Frame: Day 5: 24 hours
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Fosfomycin - 3 Doses QoD | Fosfomycin - 7 Doses QD
Number analyzed (Participants) | 18 | 18
mg/L
  Pre-dose | 66.24 (102.59) | 314.34 (257.97)
  0-4 hours post-Dose | 642.83 (521.45) | 465.74 (266.24)
  4-8 hours post-dose | 643.93 (496.86) | 608.99 (344.54)
  8-12 hours post dose | 295.01 (272.97) | 254.75 (120.71)
  12-24 hours post dose | 169.51 (112.14) | 222.20 (167.87)

19. Secondary Outcome: Urinary Bactericidal (UBT) Titers for E. Coli ATCC BAA-2323
Description: UBT for E. Coli ATCC BAA-2323
Time Frame: 24 hours on Day 1 and Day 5
Measure: Median (Inter-Quartile Range); unit: Reciprocal Titers
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Reciprocal Titers
  Day 1, >0 to 4 hr | 4 [1 to 16] | 8 [0 to 8]
  Day 1, 4 to 8 hr | 8 [2 to 16] | 2.5 [0 to 16]
  Day 1, 8 to 12 hr | 4 [0 to 8] | 3 [1 to 8]
  Day 1, 12 to 24 hr | 2 [1 to 4] | 4 [2 to 4]
  Day 5, >0 to 4 hr | 16 [4 to 32] | 4 [2 to 8]
  Day 5, 4 to 8 hr | 8 [0 to 32] | 16 [4 to 32]
  Day 5, 8 to 12 hr | 4 [0 to 8] | 4 [1 to 8]
  Day 5, 12 to 24 hr | 4 [1 to 4] | 4 [2 to 8]

20. Secondary Outcome: Urinary Bactericidal (UBT) Titers for K. Pneumoniae ATCC 33495
Description: UBT for E.coli K. Pneumoniae ATCC 33495
Time Frame: 24 hours on Day 1 and Day 5
Measure: Median (Inter-Quartile Range); unit: Reciprocal Titers
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Reciprocal Titers
  Day 1, >0 to 4 hr | 1 [0 to 2] | 0 [0 to 4]
  Day 1, 4 to 8 hr | 2 [0 to 2] | 0 [0 to 1]
  Day 1, 8 to 12 hr | 0 [0 to 0] | 0 [0 to 0]
  Day 1, 12 to 24 hr | 0 [0 to 1] | 1 [0 to 2]
  Day 5, >0 to 4 hr | 2 [0 to 4] | 1.5 [0 to 2]
  Day 5, 4 to 8 hr | 1 [0 to 4] | 2 [0 to 4]
  Day 5, 8 to 12 hr | 0 [0 to 1] | 0 [0 to 0]
  Day 5, 12 to 24 hr | 0 [0 to 1] | 1.0 [0 to 1]

21. Secondary Outcome: Urinary Bactericidal (UBT) Titers for K. Pneumoniae ATCC 700603
Description: UBT for K. Pneumoniae ATCC 700603
Time Frame: 24 hours on Day 1 and Day 5
Measure: Median (Inter-Quartile Range); unit: Reciprocal Titers
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Reciprocal Titers
  Day 1, >0 to 4 hr | 1 [0 to 2] | 0 [0 to 2]
  Day 1, 4 to 8 hr | 1 [0 to 2] | 0 [0 to 0]
  Day 1, 8 to 12 hr | 0 [0 to 1] | 0 [0 to 0]
  Day 1, 12 to 24 hr | 0 [0 to 1] | 0 [0 to 0]
  Day 5, >0 to 4 hr | 1 [0 to 2] | 1 [0 to 2]
  Day 5, 4 to 8 hr | 1 [0 to 2] | 1 [0 to 2]
  Day 5, 8 to 12 hr | 0 [0 to 1] | 0 [0 to 0]
  Day 5, 12 to 24 hr | 0 [0 to 0] | 0 [0 to 0]

22. Secondary Outcome: Urinary Bactericidal (UBT) Titers for P. Mirabilis ATCC 35659
Description: UBT for P. Mirabilis ATCC 35659
Time Frame: 24 hours on Day 1 and Day 5
Measure: Median (Inter-Quartile Range); unit: Reciprocal Titers
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Reciprocal Titers
  Day 1, >0 to 4 hr | 4 [1 to 8] | 2.5 [0 to 8]
  Day 1, 4 to 8 hr | 4 [1 to 8] | 0.5 [0 to 8]
  Day 1, 8 to 12 hr | 1 [0 to 4] | 1 [0 to 4]
  Day 1, 12 to 24 hr | 1 [1 to 4] | 2 [1 to 4]
  Day 5, >0 to 4 hr | 4 [1 to 8] | 4 [0 to 8]
  Day 5, 4 to 8 hr | 2 [0 to 8] | 4 [1 to 16]
  Day 5, 8 to 12 hr | 2 [0 to 8] | 1 [0 to 4]
  Day 5, 12 to 24 hr | 1 [0 to 4] | 2 [0 to 2]

23. Secondary Outcome: Urinary Inhibitory (UIT) Titers for E. Coli ATCC 25922
Description: UIT for E.coli ATCC 25922
Time Frame: 24 hours on Day 1 and Day 5
Measure: Median (Inter-Quartile Range); unit: Reciprocal Titers
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Reciprocal Titers
  Day 1, >0 to 4 hr | 4 [1 to 16] | 8 [0 to 16]
  Day 1, 4 to 8 hr | 8 [2 to 32] | 4.5 [0 to 16]
  Day 1, 8 to 12 hr | 4 [0 to 8] | 3 [1 to 8]
  Day 1, 12 to 24 hr | 4 [1 to 8] | 6 [2 to 8]
  Day 5, >0 to 4 hr | 8 [4 to 32] | 4 [1 to 16]
  Day 5, 4 to 8 hr | 16 [0 to 32] | 12 [1 to 32]
  Day 5, 8 to 12 hr | 4 [0 to 8] | 6 [1 to 16]
  Day 5, 12 to 24 hr | 4 [1 to 8] | 4 [1 to 8]

24. Secondary Outcome: Urinary Inhibitory (UIT) Titers for E. Coli ATCC BAA-2323
Description: UIT for E. Coli ATCC BAA-2323
Time Frame: 24 hours on Day 1 and Day 5
Measure: Median (Inter-Quartile Range); unit: Reciprocal Titers
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Reciprocal Titers
  Day 1, >0 to 4 hr | 4 [1 to 16] | 8 [0 to 8]
  Day 1, 4 to 8 hr | 8 [2 to 16] | 2.5 [0 to 16]
  Day 1, 8 to 12 hr | 4 [0 to 8] | 3 [1 to 8]
  Day 1, 12 to 24 hr | 2 [1 to 4] | 4 [2 to 4]
  Day 5, >0 to 4 hr | 16 [4 to 32] | 4 [2 to 8]
  Day 5, 4 to 8 hr | 8 [0 to 32] | 16 [4 to 32]
  Day 5, 8 to 12 hr | 4 [0 to 8] | 4 [1 to 8]
  Day 5, 12 to 24 hr | 4 [1 to 4] | 4 [2 to 8]

25. Secondary Outcome: Urinary Inhibitory (UIT) Titers for K. Pneumoniae ATCC 33495
Description: UIT for E.coli K. Pneumoniae ATCC 33495
Time Frame: 24 hours on Day 1 and Day 5
Measure: Median (Inter-Quartile Range); unit: Reciprocal Titers
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Reciprocal Titers
  Day 1, >0 to 4 hr | 1 [0 to 2] | 0 [0 to 4]
  Day 1, 4 to 8 hr | 2 [0 to 2] | 0 [0 to 1]
  Day 1, 8 to 12 hr | 0 [0 to 0] | 0 [0 to 4]
  Day 1, 12 to 24 hr | 0 [0 to 1] | 1 [0 to 2]
  Day 5, >0 to 4 hr | 2 [0 to 4] | 1.5 [0 to 2]
  Day 5, 4 to 8 hr | 1 [0 to 4] | 2 [0 to 4]
  Day 5, 8 to 12 hr | 0 [0 to 1] | 0 [0 to 0]
  Day 5, 12 to 24 hr | 0 [0 to 1] | 1 [0 to 1]

26. Secondary Outcome: Urinary Inhibitory (UIT) Titers for K. Pneumoniae ATCC 700603
Description: UIT for K. Pneumoniae ATCC 700603
Time Frame: 24 hours on Day 1 and Day 5
Measure: Median (Inter-Quartile Range); unit: Reciprocal Titers
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Reciprocal Titers
  Day 1, >0 to 4 hr | 1 [0 to 2] | 0 [0 to 2]
  Day 1, 4 to 8 hr | 1 [0 to 2] | 0 [0 to 0]
  Day 1, 8 to 12 hr | 0 [0 to 1] | 0 [0 to 0]
  Day 1, 12 to 24 hr | 0 [0 to 1] | 0 [0 to 0]
  Day 5, >0 to 4 hr | 1 [0 to 2] | 1 [0 to 2]
  Day 5, 4 to 8 hr | 1 [0 to 2] | 1 [0 to 2]
  Day 5, 8 to 12 hr | 0 [0 to 1] | 0 [0 to 0]
  Day 5, 12 to 24 hr | 0 [0 to 0] | 0 [0 to 0]

27. Secondary Outcome: Urinary Inhibitory (UIT) Titers for P. Mirabilis ATCC 35659
Description: UIT for P. Mirabilis ATCC 35659
Time Frame: 24 hours on Day 1 and Day 5
Measure: Median (Inter-Quartile Range); unit: Reciprocal Titers
Arm/Group | Fosfomycin - 3 Doses QoD Regimen | Fosfomycin - 7 Doses QD Regimen
Number analyzed (Participants) | 19 | 18
Reciprocal Titers
  Day 1, >0 to 4 hr | 4 [1 to 8] | 2.5 [0 to 8]
  Day 1, 4 to 8 hr | 4 [1 to 8] | 0.5 [0 to 8]
  Day 1, 8 to 12 hr | 1 [0 to 4] | 1 [0 to 4]
  Day 1, 12 to 24 hr | 1 [1 to 4] | 2 [1 to 4]
  Day 5, >0 to 4 hr | 4 [1 to 8] | 4 [0 to 8]
  Day 5, 4 to 8 hr | 2 [0 to 8] | 4 [1 to 16]
  Day 5, 8 to 12 hr | 2 [0 to 8] | 1 [0 to 4]
  Day 5, 12 to 24 hr | 1 [0 to 4] | 2 [0 to 2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected though 60 days following the final study visit
Groups:
- Fosfomycin - 3 Doses QoD: Fosfomycin given as a 3 gm dose, every other day for 3 doses
  Fosfomycin: Broad spectrum antibiotic
Arm/Group | Fosfomycin - 3 Doses QoD | Fosfomycin - 7 Doses QD
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/18
Other Adverse Events (participants affected / at risk) | 16/19 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosfomycin - 3 Doses QoD (N=19) | Fosfomycin - 7 Doses QD (N=18)
Clostridium difficile colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosfomycin - 3 Doses QoD (N=19) | Fosfomycin - 7 Doses QD (N=18)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 16 (16)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes